CLINICAL TRIAL: NCT00852072
Title: A Randomized Trial to Identify the Optimal Approach for Management of Difficult Bile Duct Stones
Brief Title: Randomized Trial for Extraction of Difficult Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 718940
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Common Bile Duct Stones
Keywords: common bile duct stones; mechanical lithotripsy; balloon sphincteroplasty; single-operator cholangioscopy-guided laser lithotripy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-operator cholangioscopy guided laser lithotripsy (Active Comparator): Ability to clear the bile duct of all stones in one ERCP session using laser lithotripsy-based technique, including use of mechanical lithotripsy
  Interventions: Procedure: Single-operator cholangioscopy-guided laser lithotripsy
- Balloon sphincteroplasty (Active Comparator): Ability to clear the bile duct of all stones in one ERCP session using large balloon sphincteroplasty-based technique, including use of mechanical lithotripsy
  Interventions: Procedure: Balloon Sphincteroplasty

INTERVENTIONS:
Procedure: Single-operator cholangioscopy-guided laser lithotripsy — Ability to clear the bile duct of all stones in one ERCP session using laser lithotripsy-based technique, including use of mechanical lithotripsy
  Arms: Single-operator cholangioscopy guided laser lithotripsy
Procedure: Balloon Sphincteroplasty — Ability to clear the bile duct of all stones in one ERCP session using large balloon sphincteroplasty-based technique, including use of mechanical lithotripsy
  Arms: Balloon sphincteroplasty

SUMMARY:
Removal of bile duct stones can be challenging at ERCP, particularly, when the size of the stone is at least 1.2cm, and may require more than one ERCP session. Various techniques for removal of difficult bile duct stones include using a balloon to enlarge the opening of the bile duct (large balloon sphincteroplasty), mechanical lithotripsy or single-operator cholangioscopy guided laser lithotripsy techniques. There are currently no randomized trials comparing laser lithotripsy and sphincteroplasty techniques for the removal of difficult bile duct stones and the aim of this randomized trial is to determine which technique is superior in the removal of difficult bile duct stones.

DETAILED DESCRIPTION:
Stones in the common bile duct (CBD) can result in various complications including acute cholangitis, acute pancreatitis and secondary biliary cirrhosis. Bile duct stones should therefore be removed and this can be successfully achieved in 85-90% of patients with small bile duct stones using standard endoscopic techniques. This comprises endoscopic sphincterotomy whereby the duodenal sphincter at the entrance of the bile duct is cut during endoscopic retrograde cholangiopancreatography (ERCP) and subsequent removal of the stone is achieved using standard accessories such as a basket and/or extraction balloon. However, large/difficult bile duct stones (at least 12mm in size), multiple stones and those located in non-dilated bile ducts can be difficult to remove by endoscopic sphincterotomy and using only standard accessories. In such cases, the three most commonly practiced advanced maneuvers for extraction of difficult CBD stones are mechanical lithotripsy, large balloon sphincteroplasty (LBS) of the major duodenal papilla and single operator cholangioscopy-guided laser lithotripsy (SOC-LL).

Endoscopic large balloon sphincteroplasty (using CRE Wireguided Balloon Dilatation Catheter; Boston Scientific Corp., Natick, MA, USA) is a technique in which a balloon is used to dilate the papilla located at the bile duct opening by up to 20mm (depending on size of the distal CBD) after performing an endoscopic sphincterotomy. Following dilation, the stone is removed using a basket and/or extraction balloon. This technique was shown to be effective in clearing the bile duct in 50-60% of patients with difficult bile stones in whom initial endoscopic sphincterotomy was unsuccessful.

The SpyGlass Direct Visualization System (Boston Scientific Corp., Natick, MA, USA) is a single-operator cholangioscopy system, which allows direct visualization of the bile duct stone. The main advantage of this technique is that the cholangioscope can be inserted into the endoscope and then guided through the bile duct to reach the stone. A probe can then be inserted into the cholangioscope to allow the energy from laser (laser lithotripsy) to be accurately focused onto the stone to cause stone fragmentation under direct visualization. The use of SpyGlass system with laser lithotripsy has been shown to be successful in the clearance of difficult bile duct stones in 73-100% patients.

Although various methods for removal of bile duct stones exist, there have been thus far no studies directly comparing endoscopic large balloon sphincteroplasty with cholangioscopy-guided laser lithotripsy for clearance of difficult bile duct stones. The aim of this study is therefore to compare the efficiency of the single-operator cholangioscopy-directed laser lithotripsy using the SpyGlass Direct Visualization system versus endoscopic large balloon sphincteroplasty for clearance of difficult bile duct stones.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Common bile duct stones that measure at least 1.2 cm who have failed stone removal using standard techniques at ERCP

Exclusion Criteria:

* Patients unable to provide informed consent due to any diminished capacity
* Pregnant patients or age < 18 years or prisoners
* Presence of bleeding disorders
* Patients with altered post-surgical anatomy
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment success defined as the ability to clear the bile duct of all stones in one ERCP session using either the single-operator cholangioscopy-guided laser lithotripsy-based technique or large balloon sphincteroplasty-based technique | 24 months
  Treatment success defined as the ability to clear the bile duct of all stones in one ERCP session

SECONDARY OUTCOMES:
Compare the safety of large balloon sphincteroplasty and single-operator cholangioscopy-guided laser lithotripsy techniques | 24 months
  Safety is defined as the incidence of adverse events
Compare the costs of large balloon sphincteroplasty and single-operator cholangioscopy-guided laser lithotripsy techniques | 24 months
  Costs include total costs pertaining to the treatment of bile duct stones including costs of procedure, medications, hospitalization, radiology, laboratory, anesthesia and supplies.
Compare the need for repeat interventions in large balloon sphincteroplasty and single-operator cholangioscopy-guided laser lithotripsy techniques | 24 months
  Repeat interventions is defined as the need for more than one ERCP session for complete clearance of the bile duct of stones

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript will be developed when the study is complete.

REFERENCES:
- [Derived] Bang JY, Sutton B, Navaneethan U, Hawes R, Varadarajulu S. Efficacy of Single-Operator Cholangioscopy-Guided Lithotripsy Compared With Large Balloon Sphincteroplasty in Management of Difficult Bile Duct Stones in a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Sep;18(10):2349-2356.e3. doi: 10.1016/j.cgh.2020.02.003. Epub 2020 Feb 10. PMID 32057976